CLINICAL TRIAL: NCT02416115
Title: Anti Emetic Efficacy of Combination of Ramosetron and Premixture of Naloxone With Patient-controlled Analgesia After Gynecologic Surgery
Brief Title: Anti Emetic Efficacy of Combination of Ramosetron and Premixture of Naloxone With Patient-controlled Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KNUMC-14-1037
Record Dates: First submitted 2015-04-07; First posted 2015-04-14 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2014-04

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; ramosetron; naloxone
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron; Naloxone; Sodium Chloride; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- R group (Active Comparator): Thirty minutes before end of surgery, patients in R group (n=30) received 0.3 mg ramosetron. In the post anesthetic care unit, patients in R group received PCA morphine 1 mg/ml
  Interventions: Drug: Ramosetron; Drug: Morphine
- N group (Active Comparator): Thirty minutes before end of surgery, patients in N group (n=30) received normal saline. In the post anesthetic care unit, group N received PCA mixture of naloxone 1μg/ml and morphine 1 mg/ml.
  Interventions: Drug: Naloxone; Drug: saline; Drug: Morphine
- RN group (Experimental): Thirty minutes before end of surgery, patients in Ramosetron and naloxone (RN) group (n=30) received 0.3 mg ramosetron. In the post anesthetic care unit, group RN received PCA mixture of naloxone 1μg/ml and morphine 1 mg/ml.
  Interventions: Drug: Ramosetron; Drug: Naloxone; Drug: Morphine

INTERVENTIONS:
Drug: Ramosetron — Ramosetron was given iv.
  Arms: R group; RN group
Drug: Naloxone — Naloxone added to PCA was given iv.
  Arms: N group; RN group
Drug: saline — Saline was given iv.
  Arms: N group
Drug: Morphine — Morphine in the PCA was given iv.

SUMMARY:
Postoperative nausea and vomiting (PONV) is one of the most undesirable complications after general anesthesia, and may lead to increased hospital stay and health care costs. The risk factors for PONV include sex (female population), nonsmoking status, past history of motion sickness and/or previous PONV, duration of anesthesia and surgical type (particular gynecologic surgery) and postoperative use of opioids. The overall incidence of PONV has been reported to be 30% with considerable variability, but can increase up to 69%- 80% in women undergoing gynecologic surgery with general anesthesia and morphine-patient controlled analgesia (PCA). Serotonin receptor antagonists (5-HT3) have been suggested one of the first line therapies for preventing PONV because of their efficacy and few side effects compared with other antiemetics. However, despite the use of this treatment, the incidence of PONV has been reported to be between 48 % and 50%. Naloxone is a drug used to counter the effects of opioid. It was found that administration of low dose naloxone prevents opioid side effects such as nausea and pruritus without affecting analgesia or opioid requirements in patient receiving morphine PCA. It was reported that the use of two antiemetic acting at different mechanisms is better to prevent PONV than monotherapy.

Therefore, this prospective, randomized, controlled study was designed to investigate the antiemetic efficacy of combination of ramosetron and premixture of naloxone with morphine PCA after gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking women (ASA physical status of I or II) scheduled for gynecologic surgery under general anesthesia and postoperative analgesia with a PCA device were included

Exclusion Criteria:

* known hypersensitivity to study medication; the use of antiemetics within 24 hours before surgery; the presence of gastrointestinal, renal, hepatic, or psychiatric disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The number of participants with postoperative nausea and vomiting | 24 hours
  The number of participants with postoperative nausea and vomiting